CLINICAL TRIAL: NCT00735852
Title: A Prospective Single Centre, Single Arm, Open Label Study of the Long Term Use of a LHRA Agonist (Decapeptyl SR, 11.25mg) in Combination With Livial Add Back Therapy in the Management of Chronic Cyclical Pelvic Pain in Pre Menopausal Women
Brief Title: Decapeptyl SR With Livial Add Back Therapy in the Management of Chronic Cyclical Pelvic Pain in Pre Menopausal Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STH 14404
Record Dates: First submitted 2008-08-14; First posted 2008-08-15 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Endometriosis
Keywords: endometriosis; chronic cyclical pelvic pain
MeSH Terms: conditions — Endometriosis | interventions — Triptorelin Pamoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Decapeptyl SR 11.25mg — 11.25 mgs, Intra muscular (IM) every 3 months for 2 years
  Other Names: Triptorelin acetate

SUMMARY:
This is a single-centre, open-label, within patient comparison study to assess the efficacy and safety of Decapeptyl SR when administered in combination with Livial for the treatment of women with chronic cyclical pelvic pain. This will be for a 2 year period with a 6 month post treatment follow up. The study aims to recruit 40 patients.

DETAILED DESCRIPTION:
A screening visit,will be performed and written informed consent will be obtained from the patient. In addition the patient's medical history will be checked, vital signs recorded, pain and general health questionnaires completed, blood samples collected and any prior or concomitant medications will be noted. Bone density will be determined using a DEXA scan performed in the interval between the screening and baseline visits. One month after the screening visit, patients will return to the clinic for the baseline visit. At this visit a physical examination and urine pregnancy test will be performed, vital signs measured, specific validated questionnaires on pain and endometriosis related health will be completed and symptoms of oestrogen deficiency will be documented. Patients who are still considered to be eligible for the trial will receive an injection of Decapeptyl SR 11.25 mg, and will be dispensed sufficient Livial 2.5 mg tablets to last until the next study visit. Patients will return for repeat Decapeptyl SR injections every 3 months until Month 21 at which time the last Decapeptyl SR injection will be administered. At these visits patients will also be dispensed further supplies of Livial.

Follow-up assessments will be performed during the treatment period 3, 6, 12, 18 and 24 months after the baseline visit. A final follow-up assessment will be conducted 6 months after stopping treatment. At each follow-up visit specific validated questionnaires on pain and endometriosis related health will be collected and symptoms of oestrogen deficiency will be noted. Physical examination, vital signs, bone density assessment and haematology and biochemistry analysis will be repeated at selected timepoints.

Health economic data will be collected at all study visits.

ELIGIBILITY:
Inclusion Criteria:

* aged between 18 and 45 years inclusive
* have a clinical diagnosis of chronic cyclical pelvic pain of at least 6 months duration (with or without evidence of endometriosis)
* have had investigations for possible endometriosis within three years prior to screening visit
* had regular menstrual cycles (24-42 days) for 3 months prior to screening
* treatment with LHRHa is indicated
* must be able to understand and be willing to comply with the requirements of the protocol

Exclusion Criteria:

* treated with any LHRHa within 6 months prior to screening
* treated with danazol, gestrinone or cyproterone acetate within 6 months prior to screening
* used cyclical progesterones or combined oral contraceptives within one full menstrual cycle prior to screening
* treated with any other medication other than analgesics within 3 months prior to screening
* continuous or acyclical pelvic pain
* known metabolic bone disease
* abnormal full blood count or liver or renal function at screening or within 6 months
* unexplained vaginal bleeding
* bone mineral density age adjusted T Score of -2 or below at screening visit.
* any other medical condition or abnormality that would impact on the safety or efficacy of the study treatment
* receiving treatment with coumarin or indanedione derivatives
* known contraindication or allergy or hypersensitivity to test compounds
* pregnancy or lactation
* planning a pregnancy within 31 months of screening
* of child bearing potential and unwilling to use adequate barrier contraception for the duration of the study
* received any investigational drug therapy within 30 days prior to the study
* has previously entered the study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2008-12; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
To assess the impact of treatment with Decapeptyl SR plus Livial on CCPP throughout the 24 month treatment period | baseline, month 12, month 24 and month 30

SECONDARY OUTCOMES:
To asses effect of Decapeptyl SR on pain, disability, overall health status and quality of life | baseline and 3 monthly until study end

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa Metwally, Mr, Principal Investigator — Sheffield Teaching Hopsitals Trust
Locations (1):
- Academic Unit of Reproductive and Developmental Medicine, Jessop Wing, Tree Root Walk, Sheffield, South Yorkshire, United Kingdom

REFERENCES:
- [Derived] Alshehre SM, Duffy S, Jones G, Ledger WL, Metwally M. A prospective, single-centre, single-arm, open label study of the long term use of a gonadotropin releasing hormone agonist (Triptorelin SR, 11.25 mg) in combination with Tibolone add-back therapy in the management of chronic cyclical pelvic pain. Reprod Biol Endocrinol. 2020 Apr 14;18(1):28. doi: 10.1186/s12958-020-00586-z. PMID 32290838